CLINICAL TRIAL: NCT01743482
Title: Phase II Study of Single-agent Pazopanib (Votrient®) for Patients With Relapsed or Refractory Germ-cell Tumors (GCT).
Brief Title: Pazopanib in Advanced and Cisplatin-resistant Germ Cell Tumors
Acronym: Pazotest-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Andrea Necchi, Faculty, Department of Medical Oncology, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT123/12
Record Dates: First submitted 2012-12-03; First posted 2012-12-06 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Germ Cell Tumors; Measurable Disease
Keywords: Testicular Cancer; Germ Cell Tumors; Salvage Therapy; Pazopanib
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal; Testicular Neoplasms | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pazopanib (Experimental): Patients will receive pazopanib at the dose of 800 mg/day orally until disease progression or evidence of unacceptable toxicity/side effects. The study will be performed according to Simon's two-stage optimal design.
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib
  Other Names: Votrient

SUMMARY:
This is an open label, single arm, single center, phase 2 study with the use of the antiangiogenic multikinase inhibitor pazopanib in a population of patients with germ cell tumors who are not cured following first or subsequent chemotherapy lines for metastatic disease, followed by eventual surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male gender.
* Confirmation of GCT histology based on pathologic review at Fondazione INT Milan.
* Unequivocal progression of measurable disease.
* A minimum of 2 and a maximum of 3 platinum-based chemotherapy lines for metastatic disease.
* First-line therapy should consist of at least 3 cycles of cisplatin-based chemotherapy.
* Prior single, tandem or triple high-dose chemotherapy course given as front-line or salvage therapy is allowed.

Exclusion Criteria:

* Failure to meet any of the above inclusion criteria.
* Concurrent treatment with other cytotoxic drugs or targeted therapies.
* Prior radiation therapy within 14 days of trial start.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-05-17 (Actual); Primary Completion 2016-07-27 (Actual); Study Completion 2016-07-27 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 3-months
  To evaluate the proportion of patients who are progression-free after 3 months of pazopanib.

SECONDARY OUTCOMES:
Safety and tolerability of pazopanib according to the Common Terminology Criteria for Adverse Events version 4.03 | 3 months
Response Rate | 3 months
  A response rate will be considered as the sum of complete (CR) and partial responses (PR) according to the response evaluation criteria in solid tumors (RECIST), version 1.1
Overall survival (OS) | 6 months
  OS time will be calculated as the interval from treatment start date to the date of death for any cause, with censoring at the date of last contact for patients alive. The Kaplan-Meier method will be used to estimate the OS curve.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Mi, Italy